CLINICAL TRIAL: NCT03151759
Title: Effect of Long and Short Radiotherapy on MMP-7 Levels in Rectal Cancer Treatment
Brief Title: MMP-7 Modulation by Short and Long Term Radiotherapy in Rectal Cancer Patients
Acronym: MMP-7
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: LU155-01
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No radiotherapy: Surgery only
- 25 Gray radiotherapy: Surgery after short term radiotherapy
  Interventions: Radiation: Neoadjuvant radiotherapy
- 50 Gray radiotherapy: Surgery after long term radiotherapy
  Interventions: Radiation: Neoadjuvant radiotherapy

INTERVENTIONS:
Radiation: Neoadjuvant radiotherapy — Neoadjuvant radiotherapy prior to rectal cancer surgery
  Groups: 25 Gray radiotherapy; 50 Gray radiotherapy

SUMMARY:
To analyse the effects of radiation therapy on inflammation and matrilysin levels in rectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

Adenocarcinoma of the rectum, ability to understand written and oral information, written consent.

Exclusion Criteria:

Colon cancer, benign tumors, impaired general condition of patient, declining to participate in the study, synchronous colonic tumors, logistical reasons, inability to understand written and/or oral information, previous pelvic irradiation, ongoing immunosuppressive therapy, diabetes with systemic complications.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Rectal cancer patients undergoing surgery with or without neoadjuvant radiotherapy
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2002-11-06 (Actual); Primary Completion 2007-03-16 (Actual); Study Completion 2007-03-16 (Actual)

PRIMARY OUTCOMES:
Matrilysin levels | 1 - 6 weeks
  Inflammatory markers

IPD SHARING:
Plan to Share IPD: No